CLINICAL TRIAL: NCT02673619
Title: A Phase 2a Study to Evaluate the Clinical Effect, Pharmacokinetics, Safety and Tolerability of Topically Applied Umeclidinium in Subjects With Primary Palmar Hyperhidrosis
Brief Title: A Study to Evaluate Clinical Effect, Pharmacokinetics , Safety, and Tolerability of Umeclidinium in Palmar Hyperhidrosis Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201484
Record Dates: First submitted 2016-01-25; First posted 2016-02-04 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Hyperhidrosis
Keywords: Topical; Palmar Hyperhidrosis; Umeclidinium
MeSH Terms: conditions — Hyperhidrosis | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium once daily (QD) 1.85% (Experimental): Subjects will apply UMEC topically once daily (2microliter [µL]/centimeter [cm]^2) to both the hands (palm and fingers) using graduated syringe at night before bedtime for 28 days. Randomization will be 4:1 (UMEC 1.85%: vehicle)
  Interventions: Drug: Umeclidinium
- Vehicle QD (Placebo Comparator): subjects will apply vehicle topical once daily (2µL/cm^2) to both the hands (palm and fingers) using graduated syringe at night before bedtime for 28 days.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Umeclidinium — Umeclidinium (GSK573719) 1.85% will be supplied as a clear, colourless solution, free from visible particulates, for topical application. Each subject total daily dose will be calculated as per study reference manual (SRM) using subject's hand area. A single dose of study treatment will be based on the size of the subject's hand in order to provide coverage of approximately 2µL/ cm^2. If certain pre-specified criteria for safety and tolerability are met, consideration will be given to decreasing the dose by decreasing the concentration of the topical formulation to 1.15% for the remaining subjects.
  Arms: Umeclidinium once daily (QD) 1.85%
Drug: Vehicle — The vehicle will be supplied as a clear, colorless solution, free from visible particulates, for topical application.This formulation will be similar to the umeclidinium formulation except that it will be devoid of the umeclidinium parent. A single dose of study treatment will be based on the size of the subject's hand in order to provide coverage of approximately 2µL/ cm^2
  Arms: Vehicle QD

SUMMARY:
Umeclidinium (UMEC) is a potent pan-active long-acting muscarinic antagonist (LAMA). It is anticipated that topical administration of UMEC will block stimulation of muscarinic receptors, thereby reducing the overproduction of sweat in subjects who suffer from hyperhidrosis. This study will assess the clinical effect, pharmacokinetics, safety and tolerability of topically applied UMEC following once daily topical administration, for 28 days, to the palms, in subjects with primary palmar hyperhidrosis. The study will also investigate if topically applied UMEC, at the highest possible concentration, will decrease palmar hyperhidrosis with a systemic anticholinergic adverse event profile similar to or below that observed with inhaled administration. This is a double blind (Sponsor unblind), repeat dose, randomized, parallel group, placebo controlled study. Study will enrol up to 55 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age inclusive, at the time of signing the informed consent may be considered for enrolment. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as, Pre-menopausal females with one of the following: Documented tubal ligation or Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or Hysterectomy or Documented Bilateral Oophorectomy OR Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and for 30 days after the last dose of study medication and completion of the follow-up visit.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* The subject has a HDSS score of 3 or 4.
* The subject has a diagnosis of primary, palmar hyperhidrosis, defined as excessive, palmar sweating of at least 6 months duration without apparent cause and with at least one of the following characteristics: Positive family history of hyperhidrosis or Hyperhidrosis is bilateral and relatively symmetrical or First episode of hyperhidrosis before 25 years of age or Cessation of focal sweating during sleep.
* The subject has a Baseline/Day 1 gravimetric assessment of at least 150 mg sweat produced at rest, during a period of 5 minutes separately for each palm. (Measurements can be repeated up to two times on two different days, screening and/or Baseline/Day 1 visits, but subjects need to qualify on at least one occasion for each palm.)
* The subject agrees to avoid to use nicotine-containing products (including nicotine patches) during the treatment period
* The subject is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in protocol

Exclusion Criteria:

* The subject has an unstable or life threatening cardiac disease such as: Myocardial infarction or unstable angina in the last 6 months or Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months or New York Heart Association (NYHA) Class IV heart failure
* The subject has a diagnosis of Type 1 or Type 2 diabetes, or is receiving treatment for control of blood glucose levels.
* The subject has a diagnosis of hyperthyroidism, as confirmed by thyroid stimulating hormone (TSH), or is receiving treatment for hyperthyroidism.
* The subject has a diagnosis of narrow-angle glaucoma, urinary retention, prostatic hypertrophy or bladder neck obstruction that in the opinion of the study Investigator or Medical Monitor would prevent use of an anticholinergic.
* The subject has irritation or active infection of palm area, including sweat glands.
* The subject has a current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones that the Investigator deems clinically insignificant)
* The subject has an ALT>2xUpper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening.
* The subject has QT interval corrected for heart rate (QTc) > 450 milli second (msec) or QTc > 480 msec in subjects with Bundle Branch Block.

The QTc according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.

For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the Reporting and Analysis Plan (RAP).

* The subject has a history of allergy or hypersensitivity to anticholinergic/muscarinic receptor antagonist or any ingredient of the preparation.
* The subject has had a prior surgical procedure for palmar hyperhidrosis.
* The subject has had treatment with radiofrequency and/or microwave devices for palmar hyperhidrosis
* The subject has had botulinum toxin injections for palmar hyperhidrosis in the last year prior to Baseline/Day 1
* The subject has had treatment with iontophoresis for palmar hyperhidrosis within 4 weeks prior to Baseline/Day 1
* The subject used antiperspirant on the palms within 2 weeks of the Baseline/Day 1
* The subject is a menopausal female who has had symptoms of menopause such as sweating or flushing within 3 years of Baseline/Day 1
* The subject has used any prohibited medication within the indicated washout period
* The subject tested positive for any of the following at screening or within 3 months of the first scheduled dose of study medication: Hepatitis B surface antigen (HBsAg) and Hepatitis C antibody.
* The subject has a positive pre-study drug and/or alcohol test at screening
* The subject has a positive test for Human immunodeficiency virus (HIV) antibody at screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time periods prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). This does not apply to UMEC when a subject who participated in the 1.85% cohort participates in the 1.15% cohort
* The subject has had exposure to more than four investigational medicinal products within 12 months prior to the first dosing day.
* The subject has any other condition which, in the judgment of the Investigator, would put the subject at unacceptable risk from participation in the study (e.g., subjects with renal failure).
* The subject has clinically significant abnormalities in laboratory values which, according to the Investigator, would put the subject at undue risk due to study participation.
* The subject has abnormal findings on screening ECG deemed clinically significant by the Investigator.
* The subject is pregnant or lactating or is planning on becoming pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (5):
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, College Station, Texas
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double blind, repeat dose, randomized, parallel group, placebo controlled study to examine the clinical effect, pharmacokinetics, safety and tolerability of topically applied umeclidinium (UMEC) for 28 days, to the palms, in participants with primary palmar hyperhidrosis. The study was conducted at six centers.
Pre-assignment Details: Participants were randomized in 4:1 ratio (UMEC: vehicle) to receive UMEC 1.85 percent or vehicle in higher dose cohort and UMEC 1.15 percent or vehicle in lower dose cohort. A total of 140 participants were screened, of which 82 failed screening and 58 participants were randomized into the study.
Groups:
- Higher Dose Cohort (UMEC 1.85 Percent): Participants applied UMEC 1.85 percent solution topically once a day (2 microliter [µL]/centimeter [cm]^2) to both the hands (palm and fingers) using graduated syringe at night before bedtime for 28 days.
- Higher Dose Cohort (Vehicle); Lower Dose Cohort (Vehicle): Participants received vehicle solution applied topically once a day (2 µL/cm^2) to both the hands (palm and fingers) using graduated syringe at night before bedtime for 28 days.
- Lower Dose Cohort (UMEC 1.15 Percent): Participants received UMEC 1.15 percent solution applied topically once a day (2 µL/cm^2) to both the hands (palm and fingers) using graduated syringe at night before bedtime for 28 days.
Period: Overall Study
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Started | 20 | 5 | 26 | 7
Completed | 18 | 4 | 23 | 7
Not Completed | 2 | 1 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle) | Total
Number analyzed (Participants) | 19 | 5 | 26 | 7 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] — One participant was randomized but did not receive treatment. Population: Age has been presented in two different tables to provide total for higher and lower dose seperately
  Years
    Cohort 1.85%: number analyzed (Participants) | 19 | 5 | 0 | 0 | 24
    Cohort 1.85% | 33.9 (12.31) | 23.8 (4.09) |  |  | 31.8 (11.79)
    Cohort 1.15%: number analyzed (Participants) | 0 | 0 | 26 | 7 | 33
    Cohort 1.15% |  |  | 31.8 (10.45) | 32.6 (12.55) | 32.0 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants] — One participant was randomized but did not receive treatment
  Participants
    Female | 14 | 3 | 14 | 5 | 36
    Male | 5 | 2 | 12 | 2 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — One participant was randomized but did not receive treatment
  Participants
    Race customized: AMERICAN INDIAN OR ALASKAN NATIVE | 1 | 0 | 0 | 0 | 1
    Race customized: ASIAN (ASI)-CENTRAL/SOUTH ASI HERITAGE (HER) | 1 | 0 | 1 | 0 | 2
    Race customized: BLACK OR AFRICAN AMERICAN | 5 | 0 | 5 | 2 | 12
    Race customized: NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 1 | 0 | 1
    Race customized: WHITE (W) ARABIC/NORTH AFRICAN HER | 4 | 1 | 2 | 0 | 7
    Race customized: W-W/CAUCASIAN/EUROPEAN (EUR) HER | 8 | 4 | 16 | 5 | 33
    Race customized: MULTIPLE-W-W/CAUCASIAN/EUR HER ASI - EAST ASI HER | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Posterior Probability That the Response Rate is Greater Than 50%
Description: A response rate is defined as percentage of participants who achieved at least 30 percent decrease from Baseline in gravimetric sweat production at Day 29. Baseline was latest assessment prior to first dosing. A response rate of greater than 50 percent was considered to be clinically meaningful (greater than 50 percent of participants achieving at least 30 percent decrease from Baseline in gravimetric sweat production at Day 29). The posterior probability that response rate in sweat production is greater than 50 percent was analyzed. The evaluation was performed using Bayesian analysis, in which latest pre-dose value was used as Baseline.
Time Frame: Baseline and Day 29
Population: This analysis was based on full analysis population comprised of all participants receiving study medication and having at least 1 non-missing change from Baseline efficacy assessment at/before Day 29.This analysis assessed whether response rate in UMEC arm exceeded a threshold that would warrant further development and is not relevant for vehicle.
Measure: Number; unit: Posterior Probability
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Lower Dose Cohort (UMEC 1.15 Percent)
Number analyzed (Participants) | 19 | 26
Posterior Probability | 1 | 0.9997

2. Primary Outcome: Percentage of Participants With at Least 30 Percent Reduction From Baseline in Sweat Production at Day 29
Description: Percentage of participants at Day 29 post-treatment with at least a 30 percent reduction from Baseline in sweat production measured by gravimetry. Participants remained at rest for at least 20-30 min before the measurements in order to reduce external interference. The latest pre-dose value was considered as Baseline value. The summary of percentage of participants from both the cohorts with at least 30 percent reduction from Baseline in sweat production was presented for the average of both palms.
Time Frame: Baseline and Day 29
Population: Full Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 17 | 4 | 23 | 7
Percentage of participants | 100 | 75 | 82.6 | 57.1
Statistical Analysis 1: Comparison: Higher Dose Cohort (UMEC 1.85 Percent) vs Higher Dose Cohort (Vehicle); Test type: Other; Percentage difference = 25.0, 90% CI 2-sided [-21.1 to 75.1]
Statistical Analysis 2: Comparison: Lower Dose Cohort (UMEC 1.15 Percent) vs Lower Dose Cohort (Vehicle); Test type: Other; Percentage difference = 25.5, 90% CI 2-sided [-10.2 to 59.2]

3. Secondary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline in Sweat Production at Day 29
Description: Percentage of participants at Day 29 post-treatment with at least a 50 percent reduction from Baseline in sweat production was measured by gravimetric analysis. Participants remained at rest for at least 20-30 min before the measurements in order to reduce external interference. The latest pre-dose value was considered as Baseline value. The summary of percentage of participants from both the cohorts with at least 50 percent reduction from Baseline in sweat production was presented for the average of both palms.
Time Frame: Baseline and Day 29
Population: Full Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 17 | 4 | 23 | 7
Percentage of participants | 58.8 | 75.0 | 60.9 | 42.9
Statistical Analysis 1: Comparison: Higher Dose Cohort (UMEC 1.85 Percent) vs Higher Dose Cohort (Vehicle); Test type: Other; Percentage Difference = -16.2, 90% CI 2-sided [-59.7 to 32.0]
Statistical Analysis 2: Comparison: Lower Dose Cohort (UMEC 1.15 Percent) vs Lower Dose Cohort (Vehicle); Test type: Other; Percentage Difference = 18.0, 90% CI 2-sided [-18.8 to 52.1]

4. Secondary Outcome: Change From Baseline in Amount of Sweat Produced at Day 29
Description: The amount of sweat produced was assessed by gravimetric measurement . Participants remained at rest for at least 20-30 min before the measurements in order to reduce external interference. Baseline value was the latest assessment prior to first dosing. The latest pre-dose value was considered as Baseline value.Change from Baseline value was calculated by post-dose visit value minus Baseline value. The summary of change from Baseline in sweat production has been presented for the average of both palms.
Time Frame: Baseline and Day 29
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: Milligrams (mg)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 17 | 4 | 23 | 7
Milligrams (mg) | -129.5 (114.04) | -124.8 (358.13) | -137.5 (104.87) | -112.4 (170.11)

5. Secondary Outcome: Percentage Change From Baseline/Day1 in Amount of Sweat Produced at Day 29
Description: The amount of sweat produced was assessed by gravimetric measurement . Participants remained at rest for at least 20-30 min before the measurements in order to reduce external interference. Baseline value was the latest assessment prior to first dosing. The latest pre-dose value was considered as Baseline value. Percentage change from Baseline was calculated with post-dose visit value minus Baseline value, divided by Baseline value and multiplied by 100. The summary of percentage change from Baseline in sweat production was presented for the average of both palms.
Time Frame: Baseline and Day 29
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: Percentage change of sweat produced
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 17 | 4 | 23 | 7
Percentage change of sweat produced | -60.8 (20.80) | -13.0 (113.79) | -59.5 (26.42) | -36.8 (44.88)

6. Secondary Outcome: Number of Participants With Shift of Response in HDSS Score at Day 29
Description: The HDSS was assessed based on a score 1 to 4 .The HDSS is a 4-point scale ranging from 1 (sweating never noticeable and never interferes daily activities), 2 (sweating tolerable but sometimes interferes daily activities), 3(sweating barely tolerable and frequently interferes daily activities) and 4 (sweating intolerable and always interferes daily activities s). A shift table describing change in response in participants from 1.85 percent cohort to 1.15 percent cohort has been presented for weekly average HDSS scores.
Time Frame: Baseline and Day 29
Population: Full Analysis Population
Measure: Number; unit: Participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 17 | 4 | 23 | 7
Participants
  Score 1 to 1 | 0 | 0 | 0 | 0
  Score 1 to 2 | 0 | 0 | 0 | 0
  Score 1 to 3 | 0 | 0 | 0 | 0
  Score 1 to 4 | 0 | 0 | 0 | 0
  Score 2 to 1 | 0 | 0 | 0 | 0
  Score 2 to 2 | 0 | 0 | 1 | 1
  Score 2 to 3 | 0 | 0 | 0 | 1
  Score 2 to 4 | 0 | 0 | 0 | 0
  Score 3 to 1 | 2 | 0 | 0 | 0
  Score 3 to 2 | 4 | 0 | 7 | 2
  Score 3 to 3 | 2 | 0 | 5 | 1
  Score 3 to 4 | 0 | 0 | 0 | 0
  Score 4 to 1 | 0 | 0 | 1 | 0
  Score 4 to 2 | 5 | 1 | 4 | 1
  Score 4 to 3 | 1 | 2 | 0 | 0
  Score 4 to 4 | 3 | 1 | 5 | 1

7. Secondary Outcome: Percentage of Participants With at Least 2-point Decrease From Baseline to Day 29 in HDSS Score
Description: The HDSS was assessed based on a score 1 to 4. The HDSS is a 4-point scale ranging from 1 (sweating never noticeable and never interferes daily activities), 2 (sweating tolerable but sometimes interferes daily activities), 3 (sweating barely tolerable and frequently interferes daily activities) and 4 (sweating intolerable and always interferes daily activities). Baseline value was the latest assessment prior to first dosing. The summary of percentage of participants from both the cohorts with at least 2-point decrease from Baseline in HDDS scores was presented.
Time Frame: Baseline and Day 29
Population: Full Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 17 | 4 | 23 | 7
Percentage of participants | 41.20 | 25.0 | 21.7 | 14.3
Statistical Analysis 1: Comparison: Higher Dose Cohort (UMEC 1.85 Percent) vs Higher Dose Cohort (Vehicle); Test type: Other; Percentage Difference = 16.2, 90% CI 2-sided [-32.0 to 59.7]
Statistical Analysis 2: Comparison: Lower Dose Cohort (UMEC 1.15 Percent) vs Lower Dose Cohort (Vehicle); Test type: Other; Percentage Difference = 7.5, 90% CI 2-sided [-27.7 to 42.3]

8. Secondary Outcome: Plasma Concentration After Repeat Dosing of UMEC
Description: Blood samples were collected at indicated time points. Samples were collected at nominal times relative to the proposed time of UMEC dosing. NA represents that the values were not available for specific arm or category. The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Pre dose on Day 27 and 28; 3, 6, 9, 10, 12, 16, 24 hours post dose on Day 29; 36 and 48 hours post dose on Day 30
Population: The analysis was performed on pharmacokinetic concentration (PKCNC) Population , comprised of all participants in the Safety set for whom at least one pharmacokinetic sample was obtained and analyzed.
Measure: Mean (Standard Deviation); unit: Picogram/milliliter (pg/mL)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Lower Dose Cohort (UMEC 1.15 Percent)
Number analyzed (Participants) | 12 | 22
Picogram/milliliter (pg/mL)
  DAY 27, PREDOSE, n=2,1: number analyzed (Participants) | 2 | 1
  DAY 27, PREDOSE, n=2,1 | 27.40 (23.052) | 13.70 (NA) — Standard deviation could not be calculated for n =1.
  DAY 28, PREDOSE, n=11,20: number analyzed (Participants) | 11 | 20
  DAY 28, PREDOSE, n=11,20 | 796.88 (2632.495) | 267.19 (1176.936)
  DAY 28, 3 H, n=12,19: number analyzed (Participants) | 12 | 19
  DAY 28, 3 H, n=12,19 | 0.00 (NA) — Standard deviation could not be calculated since mean is zero. | 6.21 (10.197)
  DAY 28, 6 H, n=12,18: number analyzed (Participants) | 12 | 18
  DAY 28, 6 H, n=12,18 | 2.07 (7.159) | 10.56 (31.082)
  DAY 28, 9 H, n=12,18: number analyzed (Participants) | 12 | 18
  DAY 28, 9 H, n=12,18 | 2.88 (6.883) | 9.31 (33.097)
  DAY 28, 10 H, n=11,18: number analyzed (Participants) | 11 | 18
  DAY 28, 10 H, n=11,18 | 8.07 (26.774) | 1.54 (4.491)
  DAY 28, 12 H, n=12,18: number analyzed (Participants) | 12 | 18
  DAY 28, 12 H, n=12,18 | 11.34 (39.289) | 6.03 (25.597)
  DAY 28, 16 H, n=12,18: number analyzed (Participants) | 12 | 18
  DAY 28, 16 H, n=12,18 | 24.50 (84.870) | 2.08 (8.839)
  DAY 28, 24 H, n=12,18: number analyzed (Participants) | 12 | 18
  DAY 28, 24 H, n=12,18 | 4.28 (14.809) | 2.13 (9.027)
  DAY 28, 36 H, n=12,18: number analyzed (Participants) | 12 | 18
  DAY 28, 36 H, n=12,18 | 2.03 (7.044) | 0.93 (3.936)
  DAY 28, 48 H, n=12,16: number analyzed (Participants) | 12 | 16
  DAY 28, 48 H, n=12,16 | 0.00 (NA) — Standard deviation could not be calculated since mean is zero. | 10.94 (43.775)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Blood samples were collected to measure Cmax at Day 28. Cmax is the maximum observed concentration, determined directly from the concentration-time data. The geometric mean and geometric coefficient were presented for all log transformed Cmax values.
Time Frame: Day 28
Population: PKCNC Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Log (pg/mL)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Lower Dose Cohort (UMEC 1.15 Percent)
Number analyzed (Participants) | 9 | 18
Log (pg/mL) | 18.67 (401.89) | 10.31 (152.95)

10. Secondary Outcome: Time of the Maximum Measured Plasma Concentration (Tmax) After Repeat Dosing of UMEC
Description: Blood samples were collected to measure Tmax at indicated time-points. Tmax is the time to reach Cmax, determined directly from the concentration-time data. Mean and standard deviation has been presented for Tmax values.
Time Frame: Pre dose on Day 28; 3, 6, 9, 10, 12, 16, 24 hours post dose on Day 29; 36 and 48 hours post dose on Day 30
Population: PKCNC Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Lower Dose Cohort (UMEC 1.15 Percent)
Number analyzed (Participants) | 4 | 7
Hours | 11.10 (4.287) | 5.10 (2.905)

11. Secondary Outcome: The Terminal Plasma Elimination Rate Constant (Lambda z)
Description: Blood samples were planned to be collected to measure Lambda Z. The outcome measure was not analyzed due to lack of data availability.
Time Frame: Day 28
Population: PKCNC Population. The terminal plasma elimination rate constant could not be derived for any of the participants included in the study because of insufficient data in the elimination phase.
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: The Apparent Terminal Phase Half-life (t1/2) After Repeat Dosing of UMEC
Description: Blood samples were planned to be collected to measure t1/2. The outcome measure was not analyzed due to lack of data availability.
Time Frame: Day 28
Population: PKCNC Population. The terminal phase half-life could not be derived for any of the participants included in the study because of insufficient data in the elimination phase.
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: The Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration [AUC(0-t)] and AUC Over the Dosing Interval Tau, [AUC(0-tau)] After Repeat Dosing of UMEC
Description: Blood samples were collected to measure AUC(0-t) at indicated time-points. AUC(0-t) and AUC(0-tau) was calculated by the linear up and log down trapezoidal method. Samples were collected at nominal times relative to the proposed time of UMEC dosing. The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Pre dose on Day 28; 3, 6, 9, 10, 12, 16, 24 hours post dose on Day 29; 36 and 48 hours post dose on Day 30
Population: PKCNC Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Log (h*pg/mL)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Lower Dose Cohort (UMEC 1.15 Percent)
Number analyzed (Participants) | 12 | 22
Log (h*pg/mL)
  AUC(0-t), n=9,17: number analyzed (Participants) | 9 | 17
  AUC(0-t), n=9,17 | 39.49 (648.14) | 21.87 (222.93)
  AUC(0-tau), n=6,11: number analyzed (Participants) | 6 | 11
  AUC(0-tau), n=6,11 | 964.71 (28.87) | 859.46 (0.00)

14. Secondary Outcome: Plasma Pre-dose (Trough) Concentration at the End of the Dosing Interval (Ctau)
Description: Trough (pre-dose at the end of each dosing interval) plasma concentration (Ctau) was analyzed at indicated time-points. Trough concentration samples were used for the assessment/attainment of steady state (ss). Samples were collected at nominal times relative to the proposed time of UMEC dosing. NA represents the data was not available for specific arm or category.
Time Frame: Pre dose on Day 27 and 28; 3, 6, 9, 10, 12, 16, 24 hours post dose on Day 29; 36 and 48 hours post dose on Day 30
Population: PKCNC Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Lower Dose Cohort (UMEC 1.15 Percent)
Number analyzed (Participants) | 12 | 12
pg/mL
  DAY 27;n=2,1: number analyzed (Participants) | 2 | 1
  DAY 27;n=2,1 | 22.02 (124.80) | 13.70 (NA) — Data was not available due to insufficient number of participants.
  DAY 28;n=2,2: number analyzed (Participants) | 2 | 2
  DAY 28;n=2,2 | 525.35 (270066.06) | 636.00 (8726.20)
  DAY 29;n=1,0: number analyzed (Participants) | 1 | 0
  DAY 29;n=1,0 | 51.30 (NA) — Data was not available due to insufficient number of participants. |

15. Secondary Outcome: Population Pharmacokinetic Profile After Repeat Dosing of UMEC
Description: Population pharmacokinetic profiling was planned to characterize the population pharmacokinetics of UMEC administered topically to both palms in participants with palmar hyperhidrosis. Due to the fact that the majority of the pharmacokinetic samples were below the limit of quantitation, a population pharmacokinetic analysis could not be performed.
Time Frame: Pre dose on Day 27 and 28; 3, 6, 9, 10, 12, 16, 24 hours post dose on Day 29; 36 and 48 hours post dose on Day 30
Population: PKCNC Population
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Lower Dose Cohort (UMEC 1.15 Percent)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Participants With Adverse Event (AE) and Serious Adverse Events (SAE's)
Description: An AE was any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was defined as any untoward medical occurrence that, that results in death, life-threatening, requires hospitalization or prolongation of existing hospitalization, disability/incapacity, any a congenital anomaly/birth defect or other situations at any dose.
Time Frame: Up to Day 43
Population: This analysis was performed on safety population comprised of all participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Participants
  Any AE | 8 | 4 | 7 | 1
  Any SAE | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single measurements of 12-lead ECGs were obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals. ECG values were recorded as abnormal not clinically significant (NCS) and abnormal clinically significant (CS). The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Day 1, 15 and 29
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Participants
  Day 1; abnormal NCS; n=19,5,26,7 | 13 | 3 | 12 | 1
  Day 1; abnormal CS; n=19,5,26,7 | 0 | 0 | 0 | 0
  Day 15; abnormal NCS; n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  Day 15; abnormal NCS; n=19,4,23,7 | 12 | 2 | 9 | 1
  Day 15; abnormal CS; n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  Day 15; abnormal CS; n=19,4,23,7 | 0 | 0 | 0 | 0
  Day 29; abnormal NCS; n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Day 29; abnormal NCS; n=17,4,23,7 | 11 | 3 | 9 | 1
  Day 29; abnormal CS; n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Day 29; abnormal CS; n=17,4,23,7 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Abnormal Values of Hematological Parameters
Description: Blood samples were collected from participants for evaluation of hematology parameters by Potential Clinical Chemistry Criteria. The data was presented for only those hematology parameters for which abnormal values were found (neutrophils and hemoglobin) . During the analysis, no participant in the higher dose cohort- vehicle group, nor in the lower dose cohort (for both UMEC and vehicle groups) had abnormal hematology values that met the pre-specified criteria for potential clinical importance. Hence, the data for only higher dose cohort was presented. The measurements taken at Day 29 were presented. Participants were counted in the category for their values greater than (>) reference (ref) range high and less than (<) ref range low. The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Day 29
Population: Safety Population. This outcome measures the number of participants with abnormal values of hematological parameters, therefore, only the summary for the cohort/lab parameter with abnormal data at a certain time point was presented.
Measure: Number; unit: Participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5
Participants
  Hemoglobin; > ref. range high;n=16,3: number analyzed (Participants) | 16 | 3
  Hemoglobin; > ref. range high;n=16,3 | 0 | 0
  Hemoglobin; < ref. range low;n=16,3: number analyzed (Participants) | 16 | 3
  Hemoglobin; < ref. range low;n=16,3 | 1 | 0
  Neutrophils; > ref.range high;n=16,3: number analyzed (Participants) | 16 | 3
  Neutrophils; > ref.range high;n=16,3 | 0 | 0
  Neutrophils; < ref.range low;n=16,3: number analyzed (Participants) | 16 | 3
  Neutrophils; < ref.range low;n=16,3 | 1 | 0

19. Secondary Outcome: Number of Participants With Abnormal Values of Chemistry Parameters Assessment as a Safety Measure
Description: Blood samples were collected to analyze the abnormal clinical chemistry parameters by Potential Clinical Importance Criteria. The data was presented for only those parameters for which abnormal values were found (calcium, alanine aminotransferase [ALT]). Participants in the higher dose cohort (UMEC group) had abnormal calcium values and for ALT, the abnormal values were found in lower dose cohort (UMEC group). Hence, data was presented only for these specific cohorts. Participants were counted in the category for their values > ref range high and < ref range low. The measurements taken at Day 1, Day 15 and Day 29 were presented. The participants with data available at specified time points were represented by n=x in the category titles. "n=0" in category titles represents that the data was not available for participants in respective category or arm.
Time Frame: Day 1, 15 and 29
Population: Safety Population. This outcome measures the number of participants with abnormal values of clinical chemistry parameters, therefore, only the summary for the cohort/lab parameter with abnormal data at a certain time point was presented.
Measure: Number; unit: Participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Participants
  Calcium; Day 29; > ref. range high;n=17,4,0,0: number analyzed (Participants) | 17 | 4 | 0 | 0
  Calcium; Day 29; > ref. range high;n=17,4,0,0 | 0 | 0 |  |
  Calcium; Day 29;< ref. range low;n=17,4,0,0: number analyzed (Participants) | 17 | 4 | 0 | 0
  Calcium; Day 29;< ref. range low;n=17,4,0,0 | 2 | 0 |  |
  ALT; Day 1; > ref. range high;n=0,0,25,6: number analyzed (Participants) | 0 | 0 | 25 | 6
  ALT; Day 1; > ref. range high;n=0,0,25,6 |  |  | 1 | 0
  ALT; Day 1; < ref. range low;n=0,0,25,6: number analyzed (Participants) | 0 | 0 | 25 | 6
  ALT; Day 1; < ref. range low;n=0,0,25,6 |  |  | 0 | 0
  ALT; Day 15; > ref. range high; n=0,0,23,7: number analyzed (Participants) | 0 | 0 | 23 | 7
  ALT; Day 15; > ref. range high; n=0,0,23,7 |  |  | 1 | 0
  ALT; Day 15; < ref. range low; n=0,0,23,7: number analyzed (Participants) | 0 | 0 | 23 | 7
  ALT; Day 15; < ref. range low; n=0,0,23,7 |  |  | 0 | 0

20. Secondary Outcome: Number of Participants With Abnormal Urine Analysis
Description: Urine sample were taken to analyze glucose and protein levels, blood and ketones body.Urinalysis analytes were measured by dipstick test. Results have been reported in a semi-quantitative manner as negative, Trace, 1+, 2+, 3+ and 4+, indicating proportional concentrations of the analyte in the urine sample. Abnormal laboratory values have been presented in the table. The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Day 1, 15 and 29
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Participants
  Day 1;Ketones;TRACE;n=19,5,25,7: number analyzed (Participants) | 19 | 5 | 25 | 7
  Day 1;Ketones;TRACE;n=19,5,25,7 | 1 | 0 | 1 | 1
  Day 1;Ketones;1+;n=19,5,25,7: number analyzed (Participants) | 19 | 5 | 25 | 7
  Day 1;Ketones;1+;n=19,5,25,7 | 0 | 0 | 1 | 0
  Day 1;Occult Blood;1+;n=19,5,25,7: number analyzed (Participants) | 19 | 5 | 25 | 7
  Day 1;Occult Blood;1+;n=19,5,25,7 | 0 | 0 | 0 | 1
  Day 1;Occult Blood;2+;n=19,5,25,7: number analyzed (Participants) | 19 | 5 | 25 | 7
  Day 1;Occult Blood;2+;n=19,5,25,7 | 0 | 0 | 1 | 1
  Day 1;Occult Blood;3+;n=19,5,25,7: number analyzed (Participants) | 19 | 5 | 25 | 7
  Day 1;Occult Blood;3+;n=19,5,25,7 | 0 | 0 | 1 | 1
  Day 1;Protein;TRACE;n=19,5,25,7: number analyzed (Participants) | 19 | 5 | 25 | 7
  Day 1;Protein;TRACE;n=19,5,25,7 | 2 | 1 | 2 | 0
  DAY 15;Ketones;TRACE;n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DAY 15;Ketones;TRACE;n=19,4,23,7 | 2 | 0 | 0 | 1
  DAY 15;Occult Blood;TRACE;n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DAY 15;Occult Blood;TRACE;n=19,4,23,7 | 0 | 0 | 1 | 0
  DAY 15;Occult Blood;2+;n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DAY 15;Occult Blood;2+;n=19,4,23,7 | 0 | 0 | 1 | 0
  DAY 15;Occult Blood;3+;n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DAY 15;Occult Blood;3+;n=19,4,23,7 | 2 | 0 | 0 | 1
  DAY 15;Protein;1+;n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DAY 15;Protein;1+;n=19,4,23,7 | 2 | 0 | 0 | 0
  DAY 15;Protein;2+;n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DAY 15;Protein;2+;n=19,4,23,7 | 1 | 0 | 0 | 0
  DAY 29;Glucose;TRACE;n=16,3,22,7: number analyzed (Participants) | 16 | 3 | 22 | 7
  DAY 29;Glucose;TRACE;n=16,3,22,7 | 0 | 0 | 1 | 0
  DAY 29;Ketones;TRACE;n=16,3,22,7: number analyzed (Participants) | 16 | 3 | 22 | 7
  DAY 29;Ketones;TRACE;n=16,3,22,7 | 0 | 0 | 1 | 1
  DAY 29;Ketones;1+;n=16,3,22,7: number analyzed (Participants) | 16 | 3 | 22 | 7
  DAY 29;Ketones;1+;n=16,3,22,7 | 1 | 0 | 0 | 0
  DAY 29;Occult Blood;1+;n=16,3,22,7: number analyzed (Participants) | 16 | 3 | 22 | 7
  DAY 29;Occult Blood;1+;n=16,3,22,7 | 0 | 0 | 2 | 0
  DAY 29;Occult Blood;2+;n=16,3,22,7: number analyzed (Participants) | 16 | 3 | 22 | 7
  DAY 29;Occult Blood;2+;n=16,3,22,7 | 1 | 0 | 1 | 1
  DAY 29;Occult Blood;3+;n=16,3,22,7: number analyzed (Participants) | 16 | 3 | 22 | 7
  DAY 29;Occult Blood;3+;n=16,3,22,7 | 1 | 0 | 0 | 1
  DAY 29;Protein;TRACE;n=16,3,22,7: number analyzed (Participants) | 16 | 3 | 22 | 7
  DAY 29;Protein;TRACE;n=16,3,22,7 | 1 | 0 | 1 | 2

21. Secondary Outcome: Change From Baseline in Body Temperature Assessment as a Safety Measure
Description: Body temperature was measured as a vital sign in seated position, after 5 min rest. Baseline value was the latest assessment prior to first dosing. Change from Baseline value was calculated by post-dose visit value minus Baseline value. The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Baseline, Day 15, 27, 28 and 29
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Celsius (C)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Celsius (C)
  DAY 15, n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DAY 15, n=19,4,23,7 | -0.11 (0.352) | -0.20 (0.294) | 0.14 (0.213) | -0.09 (0.227)
  DAY 27,n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  DAY 27,n=12,3,18,7 | -0.07 (0.287) | -0.07 (0.462) | 0.07 (0.277) | -0.14 (0.162)
  DAY 28,n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  DAY 28,n=12,3,20,7 | -0.03 (0.463) | 0.07 (0.551) | 0.05 (0.268) | -0.09 (0.146)
  DAY 29, n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  DAY 29, n=17,4,23,7 | 0.08 (0.222) | 0.15 (0.191) | -0.04 (0.334) | -0.11 (0.358)

22. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs including SBP and DBP were measured in a seated position, after 5 minutes rest. Baseline value was the latest assessment prior to first dosing. Change from Baseline value was calculated by post-dose visit value minus Baseline value. The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Baseline, Day 15, 27, 28 and 29
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimiters of mercury (mmHg)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Millimiters of mercury (mmHg)
  DBP;Day 15; n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  DBP;Day 15; n=19,4,23,7 | 1.5 (6.79) | 3.8 (5.68) | -1.0 (5.83) | 1.1 (12.40)
  DBP;Day 27; n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  DBP;Day 27; n=12,3,18,7 | -0.2 (4.75) | -2.3 (12.42) | -0.6 (11.08) | 3.3 (6.50)
  DBP;Day 28; n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  DBP;Day 28; n=12,3,20,7 | -1.8 (7.12) | 1.7 (12.58) | 2.3 (7.25) | 2.0 (7.16)
  DBP;Day 29; n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  DBP;Day 29; n=17,4,23,7 | -0.3 (5.64) | -0.5 (8.27) | 1.2 (8.41) | 1.0 (9.64)
  SBP;Day 15; n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  SBP;Day 15; n=19,4,23,7 | 1.2 (9.50) | 3.5 (5.32) | -7.0 (11.49) | 0.1 (10.22)
  SBP;Day 27; n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  SBP;Day 27; n=12,3,18,7 | 0.3 (12.41) | -9.3 (11.37) | -1.2 (11.12) | 3.0 (8.31)
  SBP;Day 28; n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  SBP;Day 28; n=12,3,20,7 | -2.9 (12.44) | -9.7 (20.21) | 0.8 (8.65) | 3.6 (10.52)
  SBP;Day 29; n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  SBP;Day 29; n=17,4,23,7 | 1.5 (8.38) | -2.0 (6.06) | 1.0 (10.65) | -2.4 (7.07)

23. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured in a seated position, after 5 minutes rest. Baseline value was the latest assessment prior to first dosing. Change from Baseline value was calculated by post-dose visit value minus Baseline value. The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Baseline, Day 15, 27, 28 and 29
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats/minute (min)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Beats/minute (min)
  Heart rate; Day15;n=19,4,23,7: number analyzed (Participants) | 19 | 4 | 23 | 7
  Heart rate; Day15;n=19,4,23,7 | 0.4 (6.57) | -3.8 (6.85) | 0.3 (6.43) | -1.7 (9.84)
  Heart rate;Day 27;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Heart rate;Day 27;n=12,3,18,7 | -1.6 (9.55) | -2.0 (4.00) | 0.2 (7.73) | 0.4 (6.68)
  Heart rate;Day 28;n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  Heart rate;Day 28;n=12,3,20,7 | 4.3 (12.32) | 1.7 (10.02) | 3.4 (9.46) | -1.1 (12.17)
  Heart rate;Day 29;n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Heart rate;Day 29;n=17,4,23,7 | -1.0 (8.05) | -1.0 (3.46) | -0.3 (10.19) | -6.3 (12.22)

24. Secondary Outcome: Change From Baseline in Weight
Description: Weight measurement was performed as a measure of safety. Baseline value was the latest assessment prior to first dosing. Change from Baseline value was calculated by post-dose visit value minus Baseline value.
Time Frame: Baseline and Up to Day 29
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 17 | 4 | 23 | 7
Kilograms (Kg) | 0.51 (1.892) | -0.10 (0.392) | 0.83 (2.919) | -2.67 (5.113)

25. Secondary Outcome: Number of Participants With Local Tolerability Assessments
Description: Skin tolerability was assessed by a 5-point tolerability scale ranging from 0 to 4; where 0 (no irritation), 1 (mild), 2 (moderate), 3 (severe) to 4 (Very Severe).The participants with data available at specified time points were represented by n=x in the category titles.
Time Frame: Day 1, 8, 15, 22, 27, 28, 29, 30, 36 and 43
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
Number analyzed (Participants) | 19 | 5 | 26 | 7
Participants
  Day 1;no irritation;n=19,5,26,7 | 19 | 5 | 26 | 7
  Day 1; mild;n=19,5,26,7 | 0 | 0 | 0 | 0
  Day 1; moderate;n=19,5,26,7 | 0 | 0 | 0 | 0
  Day 1; Severe;n=19,5,26,7 | 0 | 0 | 0 | 0
  Day 1; Very Severe;n=19,5,26,7 | 0 | 0 | 0 | 0
  Day 8 ;no irritation;n=19,4,25,7: number analyzed (Participants) | 19 | 4 | 25 | 7
  Day 8 ;no irritation;n=19,4,25,7 | 16 | 4 | 24 | 6
  Day 8 ;mild;n=19,4,25,7: number analyzed (Participants) | 19 | 4 | 25 | 7
  Day 8 ;mild;n=19,4,25,7 | 3 | 0 | 1 | 1
  Day 8 ;moderate;n=19,4,25,7: number analyzed (Participants) | 19 | 4 | 25 | 7
  Day 8 ;moderate;n=19,4,25,7 | 0 | 0 | 0 | 0
  Day 8 ;Severe;n=19,4,25,7: number analyzed (Participants) | 19 | 4 | 25 | 7
  Day 8 ;Severe;n=19,4,25,7 | 0 | 0 | 0 | 0
  Day 8 ;Very Severe;n=19,4,25,7: number analyzed (Participants) | 19 | 4 | 25 | 7
  Day 8 ;Very Severe;n=19,4,25,7 | 0 | 0 | 0 | 0
  Day15;no irritation;n=19,4,22,7: number analyzed (Participants) | 19 | 4 | 22 | 7
  Day15;no irritation;n=19,4,22,7 | 18 | 4 | 22 | 7
  Day 15 ;mild;n=19,4,22,7: number analyzed (Participants) | 19 | 4 | 22 | 7
  Day 15 ;mild;n=19,4,22,7 | 1 | 0 | 0 | 0
  Day 15 ;moderate;n=19,4,22,7: number analyzed (Participants) | 19 | 4 | 22 | 7
  Day 15 ;moderate;n=19,4,22,7 | 0 | 0 | 0 | 0
  Day 15 ;Severe;n=19,4,22,7: number analyzed (Participants) | 19 | 4 | 22 | 7
  Day 15 ;Severe;n=19,4,22,7 | 0 | 0 | 0 | 0
  Day 15 ;Very Severe;n=19,4,22,7: number analyzed (Participants) | 19 | 4 | 22 | 7
  Day 15 ;Very Severe;n=19,4,22,7 | 0 | 0 | 0 | 0
  Day 22 ;no irritation;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 22 ;no irritation;n=18,4,23,7 | 16 | 4 | 22 | 7
  Day 22 ;mild;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 22 ;mild;n=18,4,23,7 | 2 | 0 | 1 | 0
  Day 22 ;moderate;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 22 ;moderate;n=18,4,23,7 | 0 | 0 | 0 | 0
  Day 22 ;Severe;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 22 ;Severe;n=18,4,23,7 | 0 | 0 | 0 | 0
  Day 22 ;Very Severe;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 22 ;Very Severe;n=18,4,23,7 | 0 | 0 | 0 | 0
  Day 27 ;no irritation;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 27 ;no irritation;n=12,3,18,7 | 12 | 1 | 17 | 7
  Day 27 ;mild;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 27 ;mild;n=12,3,18,7 | 0 | 2 | 1 | 0
  Day 27 ;moderate;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 27 ;moderate;n=12,3,18,7 | 0 | 0 | 0 | 0
  Day 27 ;Severe;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 27 ;Severe;n=12,3,18,7 | 0 | 0 | 0 | 0
  Day 27 ;Very Severe;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 27 ;Very Severe;n=12,3,18,7 | 0 | 0 | 0 | 0
  Day 28 ;no irritation;n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  Day 28 ;no irritation;n=12,3,20,7 | 11 | 3 | 19 | 7
  Day 28 ;mild;n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  Day 28 ;mild;n=12,3,20,7 | 1 | 0 | 1 | 0
  Day 28 ;moderate;n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  Day 28 ;moderate;n=12,3,20,7 | 0 | 0 | 0 | 0
  Day 28 ;Severe;n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  Day 28 ;Severe;n=12,3,20,7 | 0 | 0 | 0 | 0
  Day 28 ;Very Severe;n=12,3,20,7: number analyzed (Participants) | 12 | 3 | 20 | 7
  Day 28 ;Very Severe;n=12,3,20,7 | 0 | 0 | 0 | 0
  Day 29 ;no irritation;n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Day 29 ;no irritation;n=17,4,23,7 | 15 | 4 | 23 | 6
  Day 29 ;mild;n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Day 29 ;mild;n=17,4,23,7 | 2 | 0 | 0 | 1
  Day 29 ;moderate;n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Day 29 ;moderate;n=17,4,23,7 | 0 | 0 | 0 | 0
  Day 29 ;Severe;n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Day 29 ;Severe;n=17,4,23,7 | 0 | 0 | 0 | 0
  Day 29 ;Very Severe;n=17,4,23,7: number analyzed (Participants) | 17 | 4 | 23 | 7
  Day 29 ;Very Severe;n=17,4,23,7 | 0 | 0 | 0 | 0
  Day 30 ;no irritation;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 30 ;no irritation;n=12,3,18,7 | 12 | 3 | 17 | 7
  Day 30 ;mild;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 30 ;mild;n=12,3,18,7 | 0 | 0 | 1 | 0
  Day 30 ;moderate;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 30 ;moderate;n=12,3,18,7 | 0 | 0 | 0 | 0
  Day 30 ;Severe;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 30 ;Severe;n=12,3,18,7 | 0 | 0 | 0 | 0
  Day 30 ;Very Severe;n=12,3,18,7: number analyzed (Participants) | 12 | 3 | 18 | 7
  Day 30 ;Very Severe;n=12,3,18,7 | 0 | 0 | 0 | 0
  Day 36; no irritation;n=18,3,23,7: number analyzed (Participants) | 18 | 3 | 23 | 7
  Day 36; no irritation;n=18,3,23,7 | 16 | 3 | 23 | 7
  Day 36 ;mild;n=18,3,23,7: number analyzed (Participants) | 18 | 3 | 23 | 7
  Day 36 ;mild;n=18,3,23,7 | 1 | 0 | 0 | 0
  Day 36 ;moderate;n=18,3,23,7: number analyzed (Participants) | 18 | 3 | 23 | 7
  Day 36 ;moderate;n=18,3,23,7 | 1 | 0 | 0 | 0
  Day 36 ;Severe;n=18,3,23,7: number analyzed (Participants) | 18 | 3 | 23 | 7
  Day 36 ;Severe;n=18,3,23,7 | 0 | 0 | 0 | 0
  Day 36 ;Very Severe;n=18,3,23,7: number analyzed (Participants) | 18 | 3 | 23 | 7
  Day 36 ;Very Severe;n=18,3,23,7 | 0 | 0 | 0 | 0
  Day 43 ;no irritation;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 43 ;no irritation;n=18,4,23,7 | 17 | 4 | 23 | 6
  Day 43 ;mild;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 43 ;mild;n=18,4,23,7 | 1 | 0 | 0 | 1
  Day 43 ;moderate;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 43 ;moderate;n=18,4,23,7 | 0 | 0 | 0 | 0
  Day 43 ;Severe;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 43 ;Severe;n=18,4,23,7 | 0 | 0 | 0 | 0
  Day 43 ;Very Severe;n=18,4,23,7: number analyzed (Participants) | 18 | 4 | 23 | 7
  Day 43 ;Very Severe;n=18,4,23,7 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the follow up (up to Day 43).
Description: AEs and SAEs were collected in safety population comprised of all participants who received study medication.
Arm/Group | Higher Dose Cohort (UMEC 1.85 Percent) | Higher Dose Cohort (Vehicle) | Lower Dose Cohort (UMEC 1.15 Percent) | Lower Dose Cohort (Vehicle)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/5 | 0/26 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/5 | 0/26 | 0/7
Other Adverse Events (participants affected / at risk) | 8/19 | 4/5 | 7/26 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Dose Cohort (UMEC 1.85 Percent) (N=19) | Higher Dose Cohort (Vehicle) (N=5) | Lower Dose Cohort (UMEC 1.15 Percent) (N=26) | Lower Dose Cohort (Vehicle) (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Administration site pruritus (General disorders) | 1 | 0 | 0 | 0
Administration site swelling (General disorders) | 1 | 0 | 0 | 0
Application site dryness (General disorders) | 1 | 0 | 0 | 0
Application site hypoaesthesia (General disorders) | 1 | 0 | 0 | 0
Application site paraesthesia (General disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 1
Neurogenic shock (Vascular disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Application site pain (General disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.